CLINICAL TRIAL: NCT03420612
Title: A Novel Intubation Discomfort Score Identifies Patients Feeling Painful During Unsedated Colonoscopy
Brief Title: Factors Associated With Pain During Unsedated Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: KY20163066-1
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Colonoscopy; Unsedated; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training: The training cohort was used to determine the influencing factors of the pain during the colonoscopy and establish the intubation discomfort score (IDS)
- validation: The validation cohort was used to verify the IDS

SUMMARY:
Colonoscopy is the gold standard in the diagnosis and treatment colorectal disease, but due to the uncomfortable or even painful procedure, a part of people unwilling to undergoing the examination and giving analgesic agents were recommended in several guidelines. However, use of analgesic agents have their own drawbacks, and nearly 70% patients felt no pain or only mild discomfort with the unsedated colonoscopy, routine administration of sedative or analgesic agents to all patients was considered as unnecessary. However, unsedated colonoscopy was thought to be an option for some but not for all, therefore a method to identify which patients at high risk for painful colonoscopy in preoperational stage is necessary.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years
* underwent unsedated colonoscopy

Exclusion Criteria:

* no bowel preparation or colon cleansing by enema only
* no need to reach cecum
* prior finding of severe colon stenosis or obstructing tumor
* history of colectomy
* unstable hemodynamics
* pregnant
* unable to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients of the training cohort were enrolled form Xijing Hospital of Digestive Diseases. The patients of the validation cohort were enrolled from the Shaanxi Second People's Hospital.
Sampling Method: Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
risk factor associated with painful colonoscopy rate | 2 hours
  Abdominal pain during the examination was evaluated by a previously validated 4-point verbal rating scale (no, slight, moderate, severe pain)[14], and moderate or severe pain during the procedure was defined as a "painful colonoscopy"

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, China